CLINICAL TRIAL: NCT02860273
Title: Exercise Capacity Testing in COPD Patients With High Flow Nasal Cannula
Brief Title: High Flow Nasal Cannula and Exercise Testing in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2728
Record Dates: First submitted 2016-03-29; First posted 2016-08-09 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2018-05

CONDITIONS: COPD
Keywords: Pulmonary Rehabilitation; COPD; High Flow Nasal Cannula; HFNC; Aerobic capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Flow Nasal Cannula Oxygen (Experimental): 1. Incremental Load Treadmill Test (ILTT) using HFNCO at 21%
  2. Constant Treadmill Load Test (CTLT) using HFNCO at 21%
  Interventions: Device: High Flow Nasal Cannula Oxygen
- Control Group (Other): 1. Incremental Load Treadmill Test (ILTT) at Room Air
  2. Constant Treadmill Load Test (CTLT) at Room Air
  Interventions: Device: Treadmill

INTERVENTIONS:
Device: High Flow Nasal Cannula Oxygen — Exercise capacity testing according to High Flow Nasal Cannula Oxygen at 21% in COPD patients involved in a Pulmonary Rehabilitation program.
  Other Names: HFNCO
  Arms: High Flow Nasal Cannula Oxygen
Device: Treadmill — Exercise capacity testing in COPD patients involved in a Pulmonary Rehabilitation Program.
  Arms: Control Group

SUMMARY:
In this study the investigators will determine whether the use of High Flow Nasal Cannula Oxygen during test enhances exercise performance in COPD patients on a treadmill.

DETAILED DESCRIPTION:
Design: interventional, crossover, randomized.

The main goal of this study is to compare the maximum speed reached in an Incremental Load Treadmill Test (ILTT) and max time tolerated in a Constant Treadmill Load Test (CTLT) while using High Flow Nasal Cannula Oxygen (HFNCO).

Patients will be evaluated through two different kinds of tests: Incremental Load Treadmill Test (ILTT) and Constant Treadmill Load Test (CTLT). Each test will be conducted two times, once using High Flow Nasal Cannula Oxygen and the other breathing room air.

In total, each patient will be evaluated four times on four different visits. The testing order will be randomized through STATA.

The following variables will be measured before, during and after each test:

Max speed reached in an Incremental load test: Km/h Max time tolerate in a Constant Load Test: in seconds Oxygen saturation: % Dyspnea: Modified Borg scale (0-10) Cardiac rate: beats per minute Respiratory rate: breaths per minute Blood pressure: mmHg Lower limbs fatigue: modified Borg scale (0-10) Global comfort according to the device used: visual analogue scale (VAS) 0-10

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable defined as four weeks without exacerbation.
* Signed Informed consent

Exclusion Criteria:

* Long term oxygen therapy (LTOT) or oxygen needs during exercise
* Any neuromuscular or cardiovascular condition that limits test performance
* Refusal to participate
* Contraindication for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Difference in Exercise capacity - Maximun Walking Time Tolerated | Baseline and 48 hs after baseline
  Difference in Maximun Walking time tolerated in a Constant Treadmill Load Test (CTLT) in seconds between HFNCO and Room air

SECONDARY OUTCOMES:
Difference in Dyspnea | Baseline and 48 hs after baseline
  Difference in dyspnea using Modified Borg Scale (0 - 10 points) between HFNCO and Room air
Difference in Cardiac Rate | Baseline and 48 hs after baseline
  Difference in Cardiac Rate (beats per minute) using a pulse oximetry between HFNCO and Room air
Difference in Oxygen Saturation | Baseline and 48 hs after baseline
  Difference in Oxygen Saturation using a pulse oximetry (SpO2) between HFNCO and Room air
Difference in Global Comfort | Baseline and 48 hs after baseline
  Difference in global comfort according to the device used with visual analogue scale (VAS) 0-10 between HFNCO and Room air
Difference in Lower Limbs Fatigue | Baseline and 48 hs after baseline
  Difference in Lower limbs fatigue using modified Borg scale (0-10) between HFNCO and Room air
Difference in Respiratory Rate | Baseline and 48 hs after baseline
  Difference in Respiratory rate in breaths per minute between HFNCO and Room air
Difference in Blood Pressure | Baseline and 48 hs after baseline
  Difference in of Blood pressure in mmHg between HFNCO and Room air
Difference in Exercise capacity - Maximun Walking Speed Reached | Baseline and 48 hs after baseline
  Difference in Maximun walking speed in km/h reached in an Incremental load treadmill test (ILTT) between HFNCO and Room air

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás NR Roux, PT-RT, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rabinovich RA, Vilaro J. Structural and functional changes of peripheral muscles in chronic obstructive pulmonary disease patients. Curr Opin Pulm Med. 2010 Mar;16(2):123-33. doi: 10.1097/MCP.0b013e328336438d. PMID 20071991
- [Result] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Result] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Result] Guell Rous MR, Diaz Lobato S, Rodriguez Trigo G, Morante Velez F, San Miguel M, Cejudo P, Ortega Ruiz F, Munoz A, Galdiz Iturri JB, Garcia A, Servera E; Sociedad Espanola de Neumologia y Cirugia Toracica (SEPAR). Pulmonary rehabilitation. Sociedad Espanola de Neumologia y Cirugia Toracica (SEPAR). Arch Bronconeumol. 2014 Aug;50(8):332-44. doi: 10.1016/j.arbres.2014.02.014. Epub 2014 May 17. English, Spanish. PMID 24845559
- [Result] Bolton CE, Blakey JD, Morgan MD; BTS Pulmonary Rehabilitation Guideline Development Group for the Standards of Care Committee for the BTS. The British Thoracic Society guideline on pulmonary rehabilitation in adults: your opinion is noted. Thorax. 2014 Apr;69(4):388-9. doi: 10.1136/thoraxjnl-2013-204754. Epub 2014 Jan 15. No abstract available. PMID 24430178
- [Result] Sivori M, Almeida M, Benzo R, Boim C, Brassesco M, Callejas O, Capparelli I, Conti E, Diaz M, Draghi J, Franco J, Gando S, Giuliano G, Guida R, Jolly E, Pessolano F, Rabinovich R, Ratto P, Rhodius E, Saadia M, Salvado A, Sobrino E, Victorio C. [New argentine consensus of respiratory rehabilitation 2008]. Medicina (B Aires). 2008;68(4):325-44. Spanish. PMID 18786894
- [Result] Patessio A, Carone M, Ioli F, Donner CF. Ventilatory and metabolic changes as a result of exercise training in COPD patients. Chest. 1992 May;101(5 Suppl):274S-278S. doi: 10.1378/chest.101.5_supplement.274s. PMID 1576849
- [Result] O'Donnell DE, D'Arsigny C, Webb KA. Effects of hyperoxia on ventilatory limitation during exercise in advanced chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Mar;163(4):892-8. doi: 10.1164/ajrccm.163.4.2007026. PMID 11282762
- [Result] Nonoyama ML, Brooks D, Lacasse Y, Guyatt GH, Goldstein RS. Oxygen therapy during exercise training in chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD005372. doi: 10.1002/14651858.CD005372.pub2. PMID 17443585
- [Result] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Result] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849
- [Result] Spoletini G, Alotaibi M, Blasi F, Hill NS. Heated Humidified High-Flow Nasal Oxygen in Adults: Mechanisms of Action and Clinical Implications. Chest. 2015 Jul;148(1):253-261. doi: 10.1378/chest.14-2871. PMID 25742321
- [Result] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Result] Hardinge M, Suntharalingam J, Wilkinson T; British Thoracic Society. Guideline update: The British Thoracic Society Guidelines on home oxygen use in adults. Thorax. 2015 Jun;70(6):589-91. doi: 10.1136/thoraxjnl-2015-206918. Epub 2015 Apr 27. PMID 25918120
- [Result] Cooper CB, Abrazado M, Legg D, Kesten S. Development and implementation of treadmill exercise testing protocols in COPD. Int J Chron Obstruct Pulmon Dis. 2010 Oct 12;5:375-85. doi: 10.2147/copd.s11153. PMID 21103404
- [Result] Marrugat J, Vila J, Pavesi M, Sanz F. [Estimation of the sample size in clinical and epidemiological investigations]. Med Clin (Barc). 1998 Sep 12;111(7):267-76. No abstract available. Spanish. PMID 9789243
- [Result] Laszlo G. Standardisation of lung function testing: helpful guidance from the ATS/ERS Task Force. Thorax. 2006 Sep;61(9):744-6. doi: 10.1136/thx.2006.061648. PMID 16936234
- [Result] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Result] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Result] ERS Task Force; Palange P, Ward SA, Carlsen KH, Casaburi R, Gallagher CG, Gosselink R, O'Donnell DE, Puente-Maestu L, Schols AM, Singh S, Whipp BJ. Recommendations on the use of exercise testing in clinical practice. Eur Respir J. 2007 Jan;29(1):185-209. doi: 10.1183/09031936.00046906. PMID 17197484
- [Result] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Result] Casaburi R, Kukafka D, Cooper CB, Witek TJ Jr, Kesten S. Improvement in exercise tolerance with the combination of tiotropium and pulmonary rehabilitation in patients with COPD. Chest. 2005 Mar;127(3):809-17. doi: 10.1378/chest.127.3.809. PMID 15764761
- [Result] O'Donnell DE. Hyperinflation, dyspnea, and exercise intolerance in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2006 Apr;3(2):180-4. doi: 10.1513/pats.200508-093DO. PMID 16565429
- [Result] O'Donnell DE, Revill SM, Webb KA. Dynamic hyperinflation and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):770-7. doi: 10.1164/ajrccm.164.5.2012122. PMID 11549531
- [Result] van 't Hul A, Kwakkel G, Gosselink R. The acute effects of noninvasive ventilatory support during exercise on exercise endurance and dyspnea in patients with chronic obstructive pulmonary disease: a systematic review. J Cardiopulm Rehabil. 2002 Jul-Aug;22(4):290-7. doi: 10.1097/00008483-200207000-00013. PMID 12202851
- See also: Global initiative for Chronic Obstructive Lung Disease. Update 2016 — http://goldcopd.org/global-strategy-diagnosis-management-prevention-copd-2016/